CLINICAL TRIAL: NCT05523193
Title: A Real World Study of Valvular Heart Disease in Jiangxi Province
Brief Title: Valvular Heart Disease in Jiangxi Province
Acronym: JXVD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xiao Huang (Other)
Responsible Party: Sponsor-Investigator, Xiao Huang, Principal Investigator, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Other Study IDs: 2022-07
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Valvular Heart Disease; Treatment Adherence and Compliance
Keywords: Valvular Heart Disease; Valvular regurgitation; Valvular stenosis; TAVI
MeSH Terms: conditions — Heart Valve Diseases; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Collect blood samples, tissues and body fluids according to the requirements of the sample bank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group: Treatment group (Formal treatment model group): Patients who agree and accept the surgical treatment recommendation (including medical and surgical treatment) enter the formal treatment model group.
  Those who have received any of the following treatments (including but not limited to) as recommended by the standardized treatment process are considered to have received the standardized treatment, otherwise, they have not.
  1. Surgical procedures: valve repair or replacement, left auricular ligation, left auricular clip.
  2. Internal surgery: transcatheter valve replacement, radiofrequency ablation of atrial fibrillation, and left heart ear occlusion.
  Interventions: Other: Formal treatment model
- Control group: Control group（Conventional treatment model group）:Patients who do not agree to enter the Formal treatment model group will automatically enter the Conventional treatment model group.

INTERVENTIONS:
Other: Formal treatment model — Formal treatment model , no further surgery or minimally invasive treatment was performed
  Groups: Treatment group

SUMMARY:
Study Title: A real-world study of valvular heart disease in Jiangxi Province

Research Objectives:

① Main objectives: To examine the current incidence of valvular heart disease in Jiangxi Province, to establish a "Formal treatment model" for patients with valvular heart disease, and to manage the collection of diagnostic, therapeutic and prognostic data on patients.

② Secondary objective: To investigate the composite of all-cause mortality, disabling stroke, permanent pacemaker implantation, and moderate or greater valve regurgitation in the "Formal treatment model" group and the "Conventional treatment model" group. The Conventional group was matched to patients who were not in the " Formal treatment model " during the same period.

Design type: a prospective, observational, real-world study (at least 1.5 years). No pre-established fixed treatment protocols, only a Formal treatment model,with all treatment choices made entirely by clinicians following relevant textbooks, expert consensus on clinical guidelines, and based on the patient's condition.

Subjects: All patients with moderate to severe heart valve disease were collected from the Second Affiliated Hospital of Nanchang University and hospitals at all levels in Jiangxi Province from September 2022 to September 2023.

DETAILED DESCRIPTION:
Summary of Research Protocol:

Study Title: A Real World Study of Valvular Heart Disease in Jiangxi Province

Research Objectives:

① Main objectives: To examine the current incidence of valvular heart disease in Jiangxi Province, to establish a "Formal treatment model" for patients with valvular heart disease, and to manage the collection of diagnostic, therapeutic and prognostic data on patients.

② Secondary objective: To investigate the composite of all-cause mortality, disabling stroke, permanent pacemaker implantation, and moderate or greater valve regurgitation in the "Formal treatment model" group and the "Conventional treatment model" group. The Conventional group was matched to patients who were not in the " Formal treatment model " during the same period.

Design type: a prospective, observational, real-world study (at least 1.5 years). No pre-established fixed treatment protocols, only a Formal treatment model,with all treatment choices made entirely by clinicians following relevant textbooks, expert consensus on clinical guidelines, and based on the patient's condition.

Subjects: All patients with moderate to severe heart valve disease were collected from the Second Affiliated Hospital of Nanchang University and hospitals at all levels in Jiangxi Province from September 2022 to September 2023.

Formal treatment model group: Patients who agree and accept the surgical treatment recommendation (including medical and surgical treatment) enter the formal treatment model group.

Those who have received any of the following treatments (including but not limited to) as recommended by the standardized treatment process are considered to have received the standardized treatment, otherwise, they have not.

1. Surgical procedures: valve repair or replacement, left auricular ligation, left auricular clip.
2. Internal surgery: transcatheter valve replacement, radiofrequency ablation of atrial fibrillation, and left heart ear occlusion.

Conventional treatment model group: Patients who do not agree to enter the Formal treatment model group will automatically enter the Conventional treatment model group.

ELIGIBILITY:
Inclusion Criteria:

* All moderate-to-severe heart valve disease, including aortic, mitral, and tricuspid valves;
* Comply with the ESC/EACTS Guidelines for the Management of Valvular Heart Disease (2021) indications for surgery for valvular heart disease;
* Understand and voluntarily sign the informed consent form

Exclusion Criteria:

* those with severe mental disorders and unable to express their will;
* those with obvious other abnormal signs, laboratory tests and clinical diseases that, in the judgment of the investigator, make them unsuitable for participation in the study;
* those who, in the judgment of the investigator, are unable to complete long-term follow-up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with moderate to severe heart valve disease were collected from the Second Affiliated Hospital of Nanchang University and hospitals at all levels in Jiangxi Province from September 2022 to September 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1052 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoints | 1 year after surgery or treatment
  all-cause mortality, disabling stroke, and incidence of cardiogenic stroke, permanent pacemaker implantation rate, and moderate or greater valve regurgitation at 1 year after surgery or discharge from treatment

SECONDARY OUTCOMES:
All-cause mortality | surgery or 30 days after treatment
  Including cardiac death and non-cardiac death
incidence of stroke | 30 days after discharge from hospital after surgery or treatment
  The incidence of stroke 30 days after discharge from hospital after surgery or treatment
rate of permanent pacemaker implantation | surgery or 30 days after treatment
  The rate of permanent pacemaker implantation after surgery or 30 days after treatment
Moderate or higher valvular regurgitation | immediately after the surgery or 30 days after discharge
  Moderate or higher valvular regurgitation after surgery or 30 days after discharge
Readmission rates for aortic stenosis and/or valve implantation-related complications | 30 days and 1 year after surgery or treatment
  Readmission rates for aortic stenosis and/or valve implantation-related complications at 30 days and 1 year after surgery or treatment
The incidence of intraoperative temporary valve size replacement | intraoperative
  including increasing or decreasing valve size
The incidence of abnormal valve position | during operation
  including valve displacement, valve embolism, and valve ectopic release
The incidence of implantation of two or more valves | during aortic valve replacement
  The incidence of implantation of two or more valves during aortic valve replacement
The Barthel index | 30 days and 1 year after surgery or treatment
  The Barthel index was used to evaluate the health status of the subjects
NYHA classification | 30 days and 1 year after discharge after surgery or treatment
  NYHA classification at 30 days and 1 year after discharge after surgery or treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Wu, President, Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cary T, Pearce J. Aortic stenosis: pathophysiology, diagnosis, and medical management of nonsurgical patients. Crit Care Nurse. 2013 Apr;33(2):58-72. doi: 10.4037/ccn2013820. PMID 23547127
- [Result] Carita P, Coppola G, Novo G, Caccamo G, Guglielmo M, Balasus F, Novo S, Castrovinci S, Moscarelli M, Fattouch K, Corrado E. Aortic stenosis: insights on pathogenesis and clinical implications. J Geriatr Cardiol. 2016 Sep;13(6):489-98. doi: 10.11909/j.issn.1671-5411.2016.06.001. PMID 27582763
- [Result] Dweck MR, Boon NA, Newby DE. Calcific aortic stenosis: a disease of the valve and the myocardium. J Am Coll Cardiol. 2012 Nov 6;60(19):1854-63. doi: 10.1016/j.jacc.2012.02.093. Epub 2012 Oct 10. PMID 23062541
- [Result] Sathyamurthy I, Alex S. Calcific aortic valve disease: is it another face of atherosclerosis? Indian Heart J. 2015 Sep-Oct;67(5):503-6. doi: 10.1016/j.ihj.2015.07.033. Epub 2015 Aug 21. PMID 26432749
- [Result] Soler-Soler J, Galve E. Worldwide perspective of valve disease. Heart. 2000 Jun;83(6):721-5. doi: 10.1136/heart.83.6.721. No abstract available. PMID 10814642

DOCUMENTS (1):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT05523193/Prot_000.pdf